CLINICAL TRIAL: NCT02120885
Title: An Effect of an Individualized Physical Activity Intervention for Gastric Cancer Patient Undergoing Minimally Invasive Gastrectomy: a Phase III, Prospective Randomized Controlled Trial
Acronym: Gastric cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-2013-0215
Record Dates: First submitted 2014-03-31; First posted 2014-04-23 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; minimally invasive gastrectomy; Physical activity intervention
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): physical activity intervention
  Interventions: Behavioral: physical activity intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: physical activity intervention — Exercise program is scheduled to be conducted in three phases. Phase I is in-hospital exercise program. This program will be conducted in hospital during 1 week after surgery. Phase II is home-exercise program that will be performed at home during 1 week after discharge. Phase III is main-exercise program that will be conducted the fitness center nearby hospital during 8 weeks after phase II program. Main-exercise program is focused on the functional recovery.
  Arms: Exercise group

SUMMARY:
Gastric cancer is a major health issue and one of the most common malignance in Korea. With the popularization of cancer screenings and increasing the average lifespan, the number of gastric cancer patients is increased. In the past, most of the research were concerned with survival and recovery after cancer surgery. However, as the medical technology had been developed and recovery rate and survival rate of cancer patients had risen, the patients wanted to return to a daily life and desire for participation for leisure. In other words, the patients who underwent surgery wants to maintain a high quality of life(QOL) level as like prior to cancer surgery.

DETAILED DESCRIPTION:
There are many reports on the effect of the exercise program after cancer surgery. In addition, exercise program was associated with improving the QOL and functional recovery, decreasing a mood of depression, maintaining a muscle mass and improving the survival rate.

However, the subject patients of previous studies were Western people. Therefore, The results were not disclosed whether the exercise program suited to the body characteristics of Korean people. Furthermore there was no exercise program studies for the gastric cancer patients.

Medical service for cancer patients care should include not only diagnosis, treatment as like surgery but efforts on enhancing the quality of life. In other words, post-management education and management program as like exercise program are necessary for the cancer patients after surgery. Thus, the investigators have done the pilot study about how to practice the exercise program and how to evaluate the effect on the recovery. Based on the result of pilot study which could identify the safety and the feasibility , the investigators would like to do a prospective randomized controlled study to prove the effect of exercise program after surgery

ELIGIBILITY:
Inclusion Criteria:

1. Early gastric cancer patients
2. Undergoing minimally invasive surgery
3. AGE: 20-70
4. ECOG: 0-1
5. A patient who did not exercise regularly for the last 6 months
6. A patient who signed the informed consent

Exclusion Criteria:

1. Pregnancy or plans to become pregnant
2. Cognitive disabilities
3. Other primary cancer history
4. History of major abdominal surgery except current surgery
5. Cardiopulmonary medical comorbidity
6. Living > 60 km from the hospital

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
QoL(quality of life) | 10 weeks after gastrectomy

SECONDARY OUTCOMES:
cardiopulmonary function test | 10 weeks after gastrectomy
vital signs reflecting of inflammation level | 10 weeks after gastrectomy
nutrition condition | 10 weeks after gastrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seodaemun-gu, Shinchondong, Seoul, South Korea